CLINICAL TRIAL: NCT00303771
Title: Randomized Study of Classic vs Simplified Leucovorin Calcium and Fluorouracil With or Without Irinotecan in Patients Aged At Least 75 Years With Advanced Colorectal Cancer
Brief Title: Combination Chemotherapy as First-Line Therapy in Treating Older Patients With Metastatic Colorectal Cancer That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000453855; FFCD-2001-02; EU-20546; AVENTIS-FFCD-2001-02; PFIZER-FFCD-2001-02
Record Dates: First submitted 2006-03-15; First posted 2006-03-17 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-05

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the rectum; stage IV rectal cancer; stage IV colon cancer; adenocarcinoma of the colon; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms; Colonic Neoplasms | interventions — Fluorouracil; Irinotecan; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- LV5FU2 classique (Active Comparator): LV5FU2 classique
  Interventions: Drug: fluorouracil; Drug: leucovorin calcium
- LV5FU2 classique + irinotécan (Experimental): LV5FU2 classique + irinotécan
  Interventions: Drug: fluorouracil; Drug: irinotecan hydrochloride; Drug: leucovorin calcium
- LV5FU2 simplifié (Active Comparator): LV5FU2 simplifié
  Interventions: Drug: fluorouracil; Drug: leucovorin calcium
- LV5FU2 simplifié+ irinotécan (Experimental): LV5FU2 simplifié + irinotécan
  Interventions: Drug: fluorouracil; Drug: irinotecan hydrochloride; Drug: leucovorin calcium

INTERVENTIONS:
Drug: fluorouracil
Drug: irinotecan hydrochloride
  Arms: LV5FU2 classique + irinotécan; LV5FU2 simplifié+ irinotécan
Drug: leucovorin calcium

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fluorouracil, leucovorin, and irinotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) in different doses or combinations may kill more tumor cells. It is not yet known which combination chemotherapy regimen is more effective in treating colorectal cancer.

PURPOSE: This randomized clinical trial is studying how well fluorouracil works together with leucovorin with or without irinotecan in treating older patients with metastatic colorectal cancer .

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the progression-free survival of elderly patients with unresectable metastatic colorectal cancer treated with 1 of 2 different chemotherapy regimens comprising fluorouracil and leucovorin calcium with vs without irinotecan hydrochloride.

Secondary

* Compare the tumor response rate and overall survival of patients treated with these regimens.
* Compare the tolerability of these regimens in these patients.
* Compare the quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter, prospective study. Patients are stratified according to participating center, gender, Karnofsky score (60-70% vs 80-90% vs 100%), associated comorbidities (Charlson Index 0 vs 1-2 vs 3+), age (75 to 79 years vs ≥ 80 years), alkaline phosphatase level (≤ 2 times normal vs > 2 times normal), and prior adjuvant chemotherapy (yes vs no). Patients are randomized to 1 of 4 treatment arms.

* Arm I: Patients receive leucovorin calcium IV over 2 hours and fluorouracil IV continuously over 22 hours on days 1 and 2.
* Arm II: Patients receive leucovorin calcium IV over 2 hours and fluorouracil IV continuously over 46 hours on days 1 and 2.
* Arm III: Patients receive leucovorin calcium and fluorouracil as in arm I and irinotecan hydrochloride IV over 90 minutes on day 1.
* Arm IV: Patients receive leucovorin calcium and fluorouracil as in arm II and irinotecan hydrochloride as in arm III.

In all arms, treatment repeats every 14 days in the absence of disease progression or unacceptable toxicity.

Patients undergo surgery within 3-10 weeks after completing chemotherapy.

Quality of life is assessed at baseline and then every 2 months thereafter.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 282 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the colon or rectum

  * Metastatic disease
  * Unresectable disease
* Measurable disease that is outside the field of prior irradiation
* No brain metastases

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Transaminases ≤ 5 times normal
* Bilirubin ≤ 1.5 times normal
* Alkaline phosphatase < 3 times normal (5 times normal if due to hepatic involvement)
* Creatinine clearance > 45 mL/min
* Life expectancy > 3 months
* No psychological, social, or geographical situation that would preclude study treatment
* No chronic diarrhea or enteropathy
* No coronary insufficiency or symptomatic cardiac disease
* No other malignancy unless curatively treated
* No contraindication to chemotherapy

PRIOR CONCURRENT THERAPY:

* At least 6 months since prior adjuvant chemotherapy for the primary tumor
* No prior extensive resection
* No other concurrent anticancer therapy

Ages: 75 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 282 (Actual)
Dates: Start 2003-06; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (survie sans progression) | 2011
  survie sans progression

SECONDARY OUTCOMES:
Overall Survival (survie globale) | 2011
  survie globale

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Mitry, MD, PhD, Study Chair — Hopital Ambroise Pare
Locations (77):
- France (77):
  - Centre Hospitalier d'Abbeville, Abbeville
  - Centre Hospitalier D'Agen, Agen
  - Centre hospitalier d'Alencon, Alençon
  - Clinique De Rochebelle, Alès
  - Centre Hospitalier Universitaire d'Amiens, Amiens
  - Centre Hospitalier d'Annecy, Annecy
  - Institut Sainte Catherine, Avignon
  - Hopital Duffaut, Avignon
  - Centre Hospitalier de Blois, Blois
  - Hopital Saint Andre, Bordeaux
  - Hopital Ambroise Pare, Boulogne-Billancourt
  - Centre Hospitalier Docteur Duchenne, Boulogne-sur-Mer
  - C.H. Bourg En Bresse, Bourg-en-Bresse
  - Centre Hospitalier Pierre Oudot, Bourgoin
  - Centre Hospitalier de Briey, Briey
  - Centre Medical de Bligny, Briis-sous-Forges
  - Centre hospitalier de Charleville Mezieres, Charleville-Mézières
  - Centre Hospitalier de Chalons-en-Champagne, Châlons-en-Champagne
  - Centre Hospitalier de Chateaubriant, Châteaubriant
  - Hopital Louis Pasteur, Colmar
  - Louis Mourier Hospital, Colombes
  - Centre Hospitalier Universitaire Henri Mondor, Créteil
  - Centre Hospitalier de Digne les Bains, Digne-les-Bains
  - Hopital Du Bocage, Dijon
  - Centre Hospitalier de Dreux, Dreux
  - Centre Hospitalier Intercommunal St. Aubin les Elbeuf, Elbeuf
  - Clinique Saint Vincent, Épernay
  - CHU de Grenoble - Hopital Michallon, Grenoble
  - Clinique Pasteur, Guilherand-Granges
  - Centre Hospitalier de Haguenau, Haguenau
  - Centre Hospitalier Departemental, La Roche-sur-Yon
  - Centre Hospitalier Universitaire de Bicetre, Le Kremlin-Bicêtre
  - Hopital Perpetuel Secours, Levallois-Perret
  - Hopital Robert Boulin, Libourne
  - Centre Hospital Universitaire Hop Huriez, Lille
  - Centre Hospital Regional Universitaire de Limoges, Limoges
  - Centre Hospitalier General, Longjumeau
  - Clinique Saint Jean, Lyon
  - Hopital Edouard Herriot - Lyon, Lyon
  - CHU de la Timone, Marseille
  - CHU Nord, Marseille
  - Centre Hospitalier de Martigues, Martigues
  - Centre Gray, Maubeuge
  - Centre Hospitalier de Meaux, Meaux
  - Centre Hospitalier General de Mont de Marsan, Mont-de-Marsan
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - CHU de Nancy - Hopitaux de Brabois, Nancy
  - Centre Hospitalier de Nevers, Nevers
  - Hopital de l'Archet CHU de Nice, Nice
  - C.H.U. de Nimes - Groupe Hospitals-Universitaire Caremeau, Nîmes
  - Centre Hospitalier d'Orange, Orange
  - Hopital d'Instruction des Armees du Val de Grace, Paris
  - Hopital Europeen Georges Pompidou, Paris
  - Hopital Bichat - Claude Bernard, Paris
  - CHU Pitie-Salpetriere, Paris
  - Hopital Cochin, Paris
  - Hopital Tenon, Paris
  - Centre Hospitalier - Pau, Pau
  - Centre Hospitalier de Perpignan, Perpignan
  - Hopital Haut Leveque, Pessac
  - Hopital Rene Dubos, Pontoise
  - CHU - Robert Debre, Reims
  - Polyclinique De Courlancy, Reims
  - Centre Eugene Marquis, Rennes
  - Centre Hospitalier Universitaire de Rouen, Rouen
  - Pole Sante Sarthe et Loir Hopital Pierre Daguet, Sablé-sur-Sarthe
  - Centre Rene Huguenin, Saint-Cloud
  - Hopital d'Instruction des Armees Begin, Saint-Mandé
  - Centre Hospitalier de Saint-Quentin, Saint-Quentin
  - Center Hospitalier de Sens, Sens
  - Hopital Foch, Suresnes
  - Centre Hospitalier Valence, Valence
  - Nouvelle Clinique Generale, Valence
  - Centre Hospitalier de Valenciennes, Valenciennes
  - Centre Hospitalier Intercommunal de la Haute-Saone, Vesoul
  - Institut Gustave Roussy, Villejuif
  - Centre Hospitalier de Vire, Vire

REFERENCES:
- [Result] Aparicio T, Jouve J, Teillet L, et al.: Geriatric factors to predict toxicity and dose-intensity reduction in FFCD 2001-02 phase III study comparing a first-line chemotherapy of LV5FU2 or FOLFIRI in treatment of metastatic colorectal cancer (mCRC) in elderly patients. [Abstract] J Clin Oncol 29 (Suppl 15): A-9111, 2011.
- [Result] Mitry E, Phelip JM, Bonnetain F, et al.: Phase III trial of chemotherapy with or without irinotecan in the front-line treatment of metastatic colorectal cancer in elderly patients (FFCD 2001-02 trial): results of a planned interim analysis. [Abstract] American Society of Clinical Oncology 2008 Gastrointestinal Cancers Symposium, 25-27 January 2008, Orlando, FL. A-281, 2008.
- [Result] Aparicio T, Lavau-Denes S, Phelip JM, Maillard E, Jouve JL, Gargot D, Gasmi M, Locher C, Adhoute X, Michel P, Khemissa F, Lecomte T, Provencal J, Breysacher G, Legoux JL, Lepere C, Charneau J, Cretin J, Chone L, Azzedine A, Bouche O, Sobhani I, Bedenne L, Mitry E; FFCD investigators. Randomized phase III trial in elderly patients comparing LV5FU2 with or without irinotecan for first-line treatment of metastatic colorectal cancer (FFCD 2001-02). Ann Oncol. 2016 Jan;27(1):121-7. doi: 10.1093/annonc/mdv491. Epub 2015 Oct 20. PMID 26487578
- [Result] Aparicio T, Jouve JL, Teillet L, Gargot D, Subtil F, Le Brun-Ly V, Cretin J, Locher C, Bouche O, Breysacher G, Charneau J, Seitz JF, Gasmi M, Stefani L, Ramdani M, Lecomte T, Mitry E. Geriatric factors predict chemotherapy feasibility: ancillary results of FFCD 2001-02 phase III study in first-line chemotherapy for metastatic colorectal cancer in elderly patients. J Clin Oncol. 2013 Apr 10;31(11):1464-70. doi: 10.1200/JCO.2012.42.9894. Epub 2013 Mar 4. PMID 23460711